CLINICAL TRIAL: NCT06089382
Title: A Phase III Trial of Sintilimab Plus Lenvatinib in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis (PVTT) After Surgical Resection
Brief Title: A Study to Evaluate Sintilimab Plus Lenvatinib as Adjuvant Therapy in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis (PVTT) After Surgical Resection
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant-02
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Programmed Cell Death 1; lysine kinase inhibitor; Immunotherapy; Adjuvant; Hepatocellular Carcinoma; Portal vein tumor thrombus,PVTT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab Plus Lenvatinib (Experimental)
  Interventions: Drug: Sintilimab; Drug: Lenvatinib
- TACE(one cycle) + active surveillance (Active Comparator)
  Interventions: Procedure: Transarterial Chemoembolization (TACE)

INTERVENTIONS:
Drug: Sintilimab — IV infusion of Sintilimab （200mg intravenously every 3 weeks for a total of 18 cycles or tumour recurrence）
  Other Names: IBI 308
  Arms: Sintilimab Plus Lenvatinib
Drug: Lenvatinib — 8mg orally once a day for 1 year
  Other Names: LENVIMA
  Arms: Sintilimab Plus Lenvatinib
Procedure: Transarterial Chemoembolization (TACE) — One cycle of TACE postoperatively
  Arms: TACE(one cycle) + active surveillance

SUMMARY:
To compare the impact on recurrence risk of adjuvant Sintilimab (a recombinant fully human anti-PD-1 monoclonal antibody) plus Lenvatinib for patients with hepatocellular carcinoma and portal vein tumor thrombus (PVTT ) after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histopathological diagnosis of HCC
* Undergone a curative resection
* Pathologically confirmed HCC with portal vein tumor thrombus (PVTT)
* Aged 18-75 years
* No previous systematic treatment and locoregional therapy for HCC prior to randomization
* No extrahepatic spread
* Full recovery from Curative resection within 4 weeks prior to randomization
* Child-Pugh: Grade A or B(7)
* ECOG-PS score: 0 or 1
* Adequate organ function

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinom or recurrent HCC
* Any preoperative treatment for HCC including local and systemic therapy
* Have received more than 1 cycle of adjuvant TACE following surgical resection
* Any acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* Known history of serious allergy to any monoclonal antibody or targeted anti-angiogenic drug
* Subjects with inadequately controlled hypertension or history of hypertensive crisis or hypertensive encephalopathy
* Active or history of autoimmune disease
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment
* Any persistent serious surgery-related complications; esophageal and/or gastric variceal bleeding within 6 months
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* Inability or refusal to comply with the treatment and monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Randomization up to approximately 36 months
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by BIRC, or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
RFS Rate at 12 and 24 Months | up to 24 months
Overall Survival (OS) | Randomization up to approximately 36 months
Adverse events (AEs) | Randomization up to approximately 36 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0
Quality of Life (QoL) Scale Score | Baseline up to 36 months
  Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Combined Global Health Status (GHS) / Quality of Life (QoL) Scale Score
Hepatocellular Carcinoma Module (EORTC QLQ-HCC18) Scale Score | Baseline up to 36 months
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30, with scores ranging from 0-100. Higher scores indicate more severe symptoms/problems. Change from baseline in the EORTC QLQ-HCC18 scale score will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China